CLINICAL TRIAL: NCT07362810
Title: The Impact of G-CSF Combined With IL-11 on Hematopoietic Reconstitution After Autologous Hematopoietic Stem Cell Transplantation
Brief Title: G-CSF Combined With IL-11 on Hematopoietic Reconstitution After Autologous Hematopoietic Stem Cell Transplantation
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhijun Bao, Director, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025K388-F251
Record Dates: First submitted 2026-01-02; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Mobilization of Hematopoietic Stem Cells (HSC) to Peripheral Blood (PB); Hematopoetic Stem Cell Transplantation; Hemato-oncologic Patients
Keywords: IL-11; mobilization; hematopoetic stem cell transplantation

STUDY DESIGN:
Intervention Model Description: random assigned, two groups, one group was the novel regimen of G-CSF plus IL-11, another one is the traditional regimen G-CSF alone.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- G-CSF+IL-11 (Experimental): rhG-CSF 5 μg/kg/day for 6 days plus rhIL-11 50 μg/kg/day for 5 days
  Interventions: Drug: G-CSF+IL-11
- G-CSF (Active Comparator): rhG-CSF 5 μg/kg/day subcutaneously for 6 days.
  Interventions: Drug: G-CSF Granulocyte-Colony Stimulating Factor

INTERVENTIONS:
Drug: G-CSF+IL-11 — rhG-CSF 5 μg/kg/day for 6 days plus rhIL-11 50 μg/kg/day for 5 days
  Arms: G-CSF+IL-11
Drug: G-CSF Granulocyte-Colony Stimulating Factor — rhG-CSF 5 μg/kg/day subcutaneously for 6 days
  Arms: G-CSF

SUMMARY:
Autologous hematopoietic stem cell transplantation(auto-HSCT) plays an important role in treating hematologic malignancies. Mobilization and collection of peripheral blood stem/progenitor cells is the key to successful autologous hematopoietic stem cell transplantation. Currently mobilization regimens are not enough in increasing the yield of megakaryocytic or erythroid stem/progenitor cells, resulting in a delay of hematopoietic reconstitution of platelets and erythrocytes. IL-11 and G-CSF have a synergistic role in mobilizing peripheral blood stem cells towards megakaryocytic or erythroid stem/progenitor cells in a preclinical study. Furthermore, a single-center, small cohort, prospective clinical study that has been completed in China(ChiCTR2500100054), which showed that after five days of mobilization, the combination of G-CSF and IL-11 significantly increased the number and proportion of functional megakaryocytic/erythroid progenitor cells in the peripheral blood mononuclear cells of patients, and also significantly shortened the time for platelet engraftment after transplantation, and also reduced the demand for red blood cell and platelet transfusions compared to G-CSF alone. A multi-center, prospective random clinical study is essential to compare the efficacy and safety of novel mobilization regimen with IL-11 plus G-CSF to G-CSF alone.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) with newly diagnosed multiple myeloma or lymphoma
* Suitable candidates for autologous hematopoietic stem cell transplantation (auto-HSCT)
* Zubrod (ECOG) performance status < 4
* Left ventricular ejection fraction (LVEF) > 40%
* No uncontrolled arrhythmia or unstable cardiac disease
* Corrected QT interval (QTc) < 470 ms
* No symptomatic pulmonary disease, with acceptable pulmonary function tests
* Serum alanine aminotransferase (ALT) < 4 × upper limit of normal (ULN)
* Total bilirubin < 2 × upper limit of normal (ULN)

Exclusion Criteria:

* Intolerance to auto-HSCT
* Prior exposure to other stem cell mobilizing agents
* Pregnancy or lactation
* Psychiatric disorders precluding participation
* Positive serology for HIV (HIV-1/2), hepatitis B, or hepatitis C

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
hematopoietic engraftment time (including granulocyte engraftment and platelet engraftment) | Data on engraftment will be collected daily from stem cell infusion (Day 0) until the occurrence of both engraftment events or up to a maximum of 100 days, whichever comes first.
  Granulocyte Engraftment Time: Defined as the number of days from stem cell infusion (Day 0) to the first of three consecutive days with an Absolute Neutrophil Count (ANC) > 0.5 × 10^9/L.
  Platelet Recovery Time: Defined as the number of days from stem cell infusion (Day 0) to the first day of seven consecutive days with a platelet count (PLT) ≥ 20 × 10^9/L without transfusion support.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Adverse events are monitored from the time of enrollment (first study intervention) through the end of the study, with an expected average follow-up of 12 months.
  AEs were evaluated according to the National Cancer Institute Common Terminology Criteria of Adverse Events, version 4.0.

SECONDARY OUTCOMES:
progression-free survival (PFS) and overall survival (OS) | PFS: From randomization to disease progression or death from any cause, whichever occurs first, through study completion, an average of 1 year. OS: From randomization to death from any cause, through study completion, an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Jiexian Ma, Principal Investigator — Huadong Hospitai, Fudan University
Locations (3):
- China (3):
  - The first affiliated hospital of Zhengzhou university, Zhengzhou, Henan
  - Huadong Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Tongji Hospital of Tongji University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 1 year after completion of this study
Access Criteria: all researchers can require the IPD and supporting information from principal investigator of the study (Email: jiexianma@hotmail.com)